CLINICAL TRIAL: NCT04469283
Title: Study of Caffeine Efficacy in ADCY5-related Dyskinesia - a Retrospective Study
Brief Title: Caffeine Efficacy in ADCY5-related Dyskinesia
Acronym: ADCY5-CAF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200193
Record Dates: First submitted 2020-06-23; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: ADCY5-related Dyskinesia
Keywords: ADCY5; dyskinesia; caffeine
MeSH Terms: conditions — Dyskinesia, Familial, with Facial Myokymia; Dyskinesias | interventions — Caffeine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- caffeine efficacy: Collection of preliminary data on caffeine efficacy on movement disorders in patients with ADCY5-related dyskinesia.
  Interventions: Other: caffeine and movement disorders

INTERVENTIONS:
Other: caffeine and movement disorders — Caffeine efficacy on movement disorders in patients with ADCY5-related dyskinesia.

SUMMARY:
Heterozygous mutations in ADCY5 induce hyperactivity of striatal adenylate cyclase type 5 (AC5), manifesting as early-onset hyperkinetic movement disorders. Numerous treatments have been tried without much efficacy thus far. Two patients from the same family reported efficacy of caffeine on paroxysmal episodes, both to prevent episodes and to reduce their duration (efficacy estimated to be around 80%), which was specific to caffeine as it was reproduced with caffeine citrate capsules. Interestingly, there is a rationale underlying this observation. Indeed, caffeine is an antagonist of adenosine A2A receptors (A2AR), which activate AC5 and are localized preferentially in striatal neurons that express dopamine receptors D2 .Caffeine therefore likely induces AC5 inhibition, and thus clinical improvement in patients with hyperactivity of this protein. This observation has been recently published in2019.

The investigators will collect preliminary data by interviewing our neurologist and neuropediatric colleagues, in France and abroad since it is a rare disease, on the effect of caffeine on motor symptoms and global clinical status in their ADCY5 patients.

DETAILED DESCRIPTION:
Heterozygous mutations in ADCY5 induce hyperactivity of striatal adenylate cyclase type 5 (AC5) manifesting as early-onset hyperkinetic movement disorders. The phenotype combines chorea, dystonia and/or myoclonus with frequent facial involvement, axial hypotonia, fluctuations and/or episodes of paroxysmal dyskinesia which can be nocturnal and/or painful, generally without intellectual deficiency, epilepsy or cerebellar syndrome . It is a very rare disease, affecting around twenty patients in France.

Scientific context of the research:

Numerous treatments have been tried without much efficacy thus far.

Scientific justification for the study:

Two patients from the same family reported efficacy of caffeine on paroxysmal episodes, both to prevent episodes and to reduce their duration (efficacy estimated to be around 80%), which was specific to caffeine as it was reproduced with caffeine citrate capsules. Interestingly there is a rationale underlying this situation. Indeed, caffeine is an antagonist of adenosine A2A receptors (A2AR), which activate AC5 and are localized preferentially in striatal neurons that express dopamine receptors D2. Caffeine therefore likely induces inhibition of AC5, and thus clinical improvement in patients with hyperactivity of this protein. This observation has been recently published in 2019 HYPOTHESIS Our hypothesis is that most patients with ADCY5-related dyskinesia respond well to caffeine.

This study is a multicentric retrospective study, which will be conducted in neurology and neuropediatric departments across the world.

Participants will be recruited by their own physician. This research will take place over 18 months in total: 12 month to collect all patients' data and 6 months to analyse data.

The number of participants will be between 5 and 20, depending on colleagues replies.

This research will take place over 18 months in total: 12 month to collect all patients' data and 6 months to analyse data.

ELIGIBILITY:
Inclusion criteria

* Proven genetic diagnosis of ADCY5-related dyskinesia
* Adults or children without age limits
* Past or present caffeine intake
* Non-opposition by the patient (adults) or the legal representatives (minors) in France, and patient information according to each country's legislation in other countries.

4.2. Exclusion criteria None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with genetically proven ADCY5-related dyskinesia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-07-15 (Estimated); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of responders to caffeine | 12 months
  the response being defined as an improvement of overall involuntary movements of 40% or more.

SECONDARY OUTCOMES:
Global improvement of involuntary movements, | 12 MONTHS
  Global change of involuntary movements ranging from 0 (no change) to 10 (disappearance of involuntary movements)
Global clinical change | 12 months
  Global clinical change ranging from 0 (no change) to 10 (normalization of the global clinical state)
Duration of paroxysmal episodes of movement disorders | 12 months
  Change of the duration of paroxysmal episodes of movement disorders with caffeine

REFERENCES:
- [Background] Meneret A, Gras D, McGovern E, Roze E. Caffeine and the Dyskinesia Related to Mutations in the ADCY5 Gene. Ann Intern Med. 2019 Sep 17;171(6):439. doi: 10.7326/L19-0038. Epub 2019 Jun 11. No abstract available. PMID 31181574